CLINICAL TRIAL: NCT03661008
Title: Paternal Involvement in Psychiatric Care of Adolescents Managed for Depression or Suicide Attempt
Acronym: EQIP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/CHU/07
Record Dates: First submitted 2017-11-24; First posted 2018-09-07 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2017-11

CONDITIONS: Psychiatric Disorder; Depression; Suicide, Attempted; Child Mental Disorder
MeSH Terms: conditions — Mental Disorders; Depression; Suicide, Attempted; Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adolescents with paternal involvement
- Adolescents without paternal involvement

SUMMARY:
Parental involvement, both quantitative and qualitative, is fundamental for a good psycho-emotional development of the child. The lack of parental involvement and especially paternal involvement significantly promotes the occurrence of behavioral disorders in children and later, in adolescence, the onset of depressive symptomatology. On the other hand, parental involvement has a protective role in the occurrence of behavioral disorders and decreases the risk of suicide attempts in adolescence. The authors of these cohort studies agree on the need for research on the identification of factors determining paternal involvement in order to organize specific prevention actions and targeted interventions to promote the involvement of fathers in psychiatric care of their adolescents.

The prevention of adolescent suicide attempts appears to be a real public health issue in Reunion Island with a suicide rate among under-35s twice as high as in Reunion than in metropolitan France.

This work is a continuation of the guidelines of good practice of the High Authority of Health (HAS) which insist on the importance of "supporting the parental function by health and public action".

ELIGIBILITY:
Inclusion Criteria:

Teenagers aged 13 to 17

* managed for a depressive episode (ADRS score> 3) or for a suicide attempt
* speaking and understanding French and / or Creole language

Exclusion Criteria:

* fathers without legal responsibility for the child
* absence of consent of the adolescent or those responsible for parental authority

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Teenagers consulting in the adolescents psychiatric unit of the University Hospital of Reunion Island
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Proportion in the most incident factors influencing paternal involvement in psychiatric care of adolescents | One hour after inclusion
  After textual analysis of the interviews (qualitative analysis)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Réunion, Saint-Pierre, Reunion Island, France

IPD SHARING:
Plan to Share IPD: No